CLINICAL TRIAL: NCT02911311
Title: Conbercept vs Panretinal Photocoagulation for the Management of Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Director of ophthalmology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONTINENT
Record Dates: First submitted 2016-09-17; First posted 2016-09-22 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: conbercept; anti-VEGF agent; panretinal photocoagulation
MeSH Terms: interventions — KH902 fusion protein; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVC group (Experimental): intravitreal injection of conbercept (IVC) group：all study eyes randomised to receive conbercept will receive an intravitreal injection of conbercept 2 mg/ 0.05 mL at baseline and at 1 and 2 moths. Further treatment since months 3 is determined by the degree of regression of neovascularization (NV) of disc and elsewhere on clinical examination
  Interventions: Drug: intravitreal injection of conbercept
- PRP group (Active Comparator): panretinal photocoagulation (PRP) group:all study eyes randomised to receive PRP will receive an fill-in PRP in 1-2 two weekly sessions as per routine clinical practice with emphasis on targeting retinal nonperfusion areas
  Interventions: Device: PRP

INTERVENTIONS:
Drug: intravitreal injection of conbercept — conbercept is an anti-VEGF agent and is approved by the Food and Drug Administration for wet age-related macular degeneration
  Other Names: KH-902 (Chengdu Kanghong Biotech Co., Ltd., Sichuan, China)
  Arms: IVC group
Device: PRP — panretinal photocoagulation (PPR) is the standard treatment for proliferative diabetic retinopathy (PDR) and is applied to the peripheral retinal tissue to ablate areas of the peripheral retina and thereby reduce retinal oxygen consumption
  Arms: PRP group

SUMMARY:
Panretinal photocoagulation (PRP) has been the standard treatment for Proliferative diabetic retinopathy (PDR) since the Diabetic Retinopathy Study demonstrated its benefit nearly 40 years ago,but PRP has inevitable adverse effects on visual function. Intravitreal injection of vascular endothelial growth factor(VEGF) can induce short-term regression of retinal neovascularization(NV). The purpose is to assess and compare the efficacy and safety between intravitreal injection of conbercept and PRP.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is a leading cause of vision loss in patients with diabetes mellitus,which of the initial manifestation of PDR is retinal neovascularization at the disc or elsewhere.Panretinal photocoagulation (PRP) has been the standard treatment for PDR since the Diabetic Retinopathy Study demonstrated its benefit nearly 40 years ago,but PRP has inevitable adverse effects on visual function including peripheral visual field defects, night vision loss, loss of contrast sensitivity.Recent evidences have indicated that anti-vascular endothelial growth factor(VEGF) treatment can reduce the severity and delay the progression of DR.However,the impact of this treatment on visual function and the effect of anti-VEGF agents on retinal neovascularization compared with PRP remain unclear. It is possible that a long-acting anti-VEGF agent such as conbercept. So we design the study with is a prospective randomized controlled trial about Intravitreal injection of conbercept versus PRP on PDR.Primary outcome is the change in BCVA from screening to 12 months in the study eye measured in the ETDRS letter score at 4 m

ELIGIBILITY:
Inclusion Criteria:

1. Participants of either sex aged 18 years or over.
2. Diagnosis of diabetes mellitus (type 1 or 2).
3. Best-corrected visual acuity (BCVA) in the study eye better than or equal to 30 Early Treatment Diabetic Retinopathy Study (ETDRS) letters
4. PDR with no evidence of previous PRP.
5. Media clarity, pupillary dilation and participant cooperation sufficient for adequate fundus photographs.

Exclusion Criteria:

1. a glycated haemoglobin (HbA1c) level of more than 10%;
2. Blood pressure > 180/100 mmHg
3. Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months
4. dialysis or renal transplant
5. Systemic anti-VEGF or pro-VEGF treatment within 6 months prior to randomization
6. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years
7. Traction retinal detachment involving the macula
8. Exam evidence of neovascularization of the angle
9. History of major ocular surgery or anticipated within the next 6 months following randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is mean visual acuity change(BCVA) | 12 months
  Primary outcome is the change in BCVA from screening to 12 moths in the study eye measured in the ETDRS letter score at 4 m

SECONDARY OUTCOMES:
Visual acuity outcomes in terms of visual gain or loss | 6 months and 12 months
  visual gain refers to the proportion of visual improvement ≥ 15 letters at 6-month follow-up, visual loss refers to the proportion of visual reduction ≤ 15 letters at 6-month and 12-month follow-up
the regression patterns of new vessels | 6 months and 12 months
  the complete regression proportion of new retinal vessels is evaluated by the fundus photography and fundus fluorescein angiography at 6 months and 12 months
proportion of patients developing macular oedema, vitreous haemorrhage and vitrectomy | 12 months
  proportion of patients developing macular oedema, vitreous haemorrhage and vitrectomy at months
change of visual field | 12 months
  change of visual field will be evaluated by the perimeter
change of retinal function | 12 months
  change of retinal function measured by electroretinography(ERG)
change of macular capillary density | 12 months
  change of macular capillary density measured by Optical coherence tomography angiography
change of central retinal thickness | 12 months
  change of central retinal thickness measured by Optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Dr., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- See also: Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial — http://www.ncbi.nlm.nih.gov/pubmed/26565927